CLINICAL TRIAL: NCT06051344
Title: Effect of Zoledronic Acid in Primary Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Effect of Zoledronic Acid in Primary Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toufiqe-E-Ealahi (Other)
Responsible Party: Sponsor-Investigator, Toufiqe-E-Ealahi, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bisphosphonate in OA
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Primary Osteoarthritis
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: . Total 92 primary knee OA patients will be enrolled by following the inclusion criteria of ages 50 years and above with primary knee OA informed written consent. Then randomization will be done into group A and group B following a randomization table, each consist of 46 patients. Consecutive sampling technique will be followed. Primary knee OA will be diagnosed on the basis of ACR clinical and radiological criteria. Relevant laboratory investigations will be done. Baseline pain status will be measured by Bangla version of Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), visual analog scale (VAS) and numerical rating scale (NRS) and quality of life will be measure by European quality of life scale (EQ-5D-5L). Then one group will receive single infusion of 5mg zoledronic acid and another group will receive the placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A, case group (Experimental): . Total 92 primary knee OA patients will be enrolled by following the inclusion criteria of ages 50 years and above with primary knee OA informed written consent. Then randomization will be done into group A and group B following a randomization table, each consist of 46 patients. Consecutive sampling technique will be followed. Primary knee OA will be diagnosed on the basis of ACR clinical and radiological criteria. Relevant laboratory investigations will be done. Baseline pain status will be measured by Bangla version of Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), visual analog scale (VAS) and numerical rating scale (NRS) and quality of life will be measure by European quality of life scale (EQ-5D-5L). Then one group will receive single infusion of 5mg zoledronic acid and another group will receive the placebo
  Interventions: Drug: Zoledronic acid
- B, control group (Experimental): . Total 92 primary knee OA patients will be enrolled by following the inclusion criteria of ages 50 years and above with primary knee OA informed written consent. Then randomization will be done into group A and group B following a randomization table, each consist of 46 patients. Consecutive sampling technique will be followed. Primary knee OA will be diagnosed on the basis of ACR clinical and radiological criteria. Relevant laboratory investigations will be done. Baseline pain status will be measured by Bangla version of Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), visual analog scale (VAS) and numerical rating scale (NRS) and quality of life will be measure by European quality of life scale (EQ-5D-5L). Then one group will receive single infusion of 5mg zoledronic acid and another group will receive the placebo
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — . Total 92 primary knee OA patients will be enrolled by following the inclusion criteria of ages 50 years and above with primary knee OA informed written consent. Then randomization will be done into group A and group B following a randomization table, each consist of 46 patients. Consecutive sampling technique will be followed. Primary knee OA will be diagnosed on the basis of ACR clinical and radiological criteria. Relevant laboratory investigations will be done. Baseline pain status will be measured by Bangla version of Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), visual analog scale (VAS) and numerical rating scale (NRS) and quality of life will be measure by European quality of life scale (EQ-5D-5L). Then one group will receive single infusion of 5mg zoledronic acid and another group will receive the placebo

SUMMARY:
We try to find out the effect of zoledronic acid over pain of primary knee osteoarthritis and also functional status in a period of 6 months.

DETAILED DESCRIPTION:
This will be a double blind placebo controlled randomized clinical trial at department of rheumatology, Bangabandhu Seikh Mujib Medical University (BSMMU) from January 2023 to December 2023. Total 92 primary knee OA patients will be enrolled by following the inclusion criteria of ages 50 years and above with primary knee OA informed written consent. Then randomization will be done into group A and group B following a randomization table, each consist of 46 patients. Consecutive sampling technique will be followed. Primary knee OA will be diagnosed on the basis of ACR clinical and radiological criteria. Relevant laboratory investigations will be done. Baseline pain status will be measured by Bangla version of Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), visual analog scale (VAS) and numerical rating scale (NRS) and quality of life will be measure by European quality of life scale (EQ-5D-5L). Then one group will receive single infusion of 5mg zoledronic acid and another group will receive the placebo. Each patient will be allowed take NSAIDs on requirement basis with documentation and follow non pharmacological treatment of OA. At the end of 6 months, again pain and functional status will be measured by WOMAC scale

ELIGIBILITY:
Inclusion Criteria:

1. >= 50 years
2. Knee OA by ACR criteria
3. Patient who will be willing to participate in the study

Exclusion Criteria:

* 1. Known inflammatory arthritis 2. BMI >= 40 kg/m2 3. Prior diagnosis of cancer 4. Prior use of bisphosphonates 5. Use of intra articular corticosteroid or hyaluronic acid preparations within 3months 6. Metabolic causes of OA (crystal associated arthritis, acromegaly, wilson's disease, haemachromatosis, Hyperparathyroidism, DM) 7. Mechanical causes of OA (epiphyseal dysplasia, congenital dislocations, limb-length inequality, hypermobility syndromes, avascular necrosis)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain status | 0,3 and 6 month
  by 1. Western Ontario McMaster Universities Osteoarthritis index Total 24 domains. Each domain range from none-0, mild-1, moderate -2, severe-3, extreme-4. Total score ranging from 0 to 96

CONTACTS AND LOCATIONS:
Overall Officials: kalam azad, FCPS MD, Study Chair — Rheumatologist
Locations (1):
- Department of rheumatology, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No